CLINICAL TRIAL: NCT06119451
Title: The Role of Traditional Music Therapy on Burnout Syndrome Among Healthcare Workers: Psycho-Neuro-Immuno-Endocrine Aspects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Yanuar Ardani, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YArdani
Record Dates: First submitted 2023-10-24; First posted 2023-11-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Burnout, Professional
Keywords: burnout syndrome; music therapy; healthcare workers; maslach burnout inventory; heart rate variability; T cell regulator; IgA; cortisol; endorphine
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: randomized control trial using pre and post test control group design¸
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Participants who will be given both educational video and traditional music therapy 3 times a week for 4 weeks in a row. This group will get Maslach Burnout Inventory, Heart Rate Variability, IgA, T cell regulator, cortisol, and endorphine score evaluated before, in the middle, right after finishing intervention, and 2 weeks after intervention.
  Interventions: Behavioral: Traditional Music Therapy
- Control group (No Intervention): Participants who will be given only educational video. This group will get Maslach Burnout Inventory, Heart Rate Variability, IgA, T cell regulator, cortisol, and endorphine score evaluated before, in the middle, right after finishing intervention, and 2 weeks after intervention.

INTERVENTIONS:
Behavioral: Traditional Music Therapy — Intervention using traditional music therapy as an alternative therapy for burnout syndrome
  Arms: Interventional Group

SUMMARY:
The goal of this clinical trial study is to learn about the role of traditional music therapy on burnout syndrome among healthcare workers, based on psychology, neurology, immunology, and endocrinology aspects. The main questions it aims to answer are :

1. How traditional music therapy can improve psychological aspects (emotional exhaustion, depersonalisation, and personal accomplishment) among healthcare workers with burnout syndrome?
2. How traditional music therapy can improve neuroautonom aspects (heart rate variability) among healthcare workers with burnout syndrome?
3. How traditional music therapy can improve immunology aspects (IgA and T cell regulator) among healthcare workers with burnout syndrome?
4. How traditional music therapy can improve endocrinology aspects (cortisol and endorphine) among healthcare workers with burnout syndrome?

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn about the role of traditional music therapy on burnout syndrome among healthcare workers. The investigators will collected about 80 participants, which eventually get divided into intervention (40 participants) and control (40 participants) group. Participants will get examined using Maslach Burnout Inventory-Human Service Survey for rating their burnout sydnrome. Before starting the intervention, both group will get assessed for their heart rate variability, IgA and T cell regulator level, and cortisol and endorphine level. After that, Intervention group will get traditional music therapy and educational video 3 session a week for about 4 weeks. And control group will only get educational video.

Both group will be assessed for their heart rate variability and their laboratory markers three times, 2 weeks after starting the intervention, right after finishing all intervention session on week 4, and 2 weeks after the intervention is done. Investigators will compare the results between control group (educational video only without any music therapy) and intervention group (traditional music therapy and educational video) to see if there are any role of traditional music therapy on burnout syndrome based on psychology-neuroautonom-immunology-endocrinology aspects.

ELIGIBILITY:
Inclusion Criteria:

* Agreed to participate in this study by signing an informed consent sheet
* Above 18 years old
* Doctors or nurses working in RSUP dr Kariadi Semarang
* MBI-HSS score show intermediate-severe burnout
* Meet the requirements for an HRV examination
* Have been working for minimum one year on each instalation

Exclusion Criteria:

* Above 60 years old
* Have history of chronic illness such as cancer, thyroid, and cardiovascular disease
* Taking drugs that affect central nervous system
* Hearing loss and disorder
* Psychosis, anxiety,depression and any other psychological disorder
* Pregnant women
* Does not like music

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Maslach Burnout Inventory Human Services Survey | one month
  an instrument developed to capture burnout for health professionals The Maslach Burnout Inventory (MBI) is a measuring tool that is generally used to assess whether you are at risk of burnout. To explain the risk of burnout, the MBI assesses three components, namely fatigue, depersonalization and self-achievement. Each statement shows a score that explains your response. Put a check mark (√) on each number that you think represents your opinion about the statement listed in the column below.
  0 : never
  1. : Several times a year
  2. : Less than or once a month
  3. : Several times a month
  4. : Once a week 5: Several times a week
  6 : Every day A participant can be categorized as burnout if he has an exhaustion score ≥ 24, a cynicism score ≥ 9, and a (reversed) accomplishment score ≥ 19.
Heart Rate Variability | one month
  Heart rate variability (HRV) is the fluctuation in the time intervals between adjacent heartbeats. HRV indexes neurocardiac function and is generated by heart-brain interactions and dynamic non-linear autonomic nervous system (ANS) processes.
Immunoglobulin A level | one month
  Evaluate Immunoglobulin A level using saliva
T cell regulator | one month
  Evaluate T cell regulator level using blood
Cortisol | one month
  Evaluate cortisol level on saliva
Endorphine | one month
  Evaluate endorphine level on saliva

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP dr. Kariadi Semarang, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Witte M, Pinho ADS, Stams GJ, Moonen X, Bos AER, van Hooren S. Music therapy for stress reduction: a systematic review and meta-analysis. Health Psychol Rev. 2022 Mar;16(1):134-159. doi: 10.1080/17437199.2020.1846580. Epub 2020 Nov 27. PMID 33176590
- [Background] Rahayu DS, Atmoko A, Muslihati M, Setyowati AJ, Mudjijanti F. Establishing Music Therapy as an Alternative to Reducing Compassion Fatigue among Health Workers. Prehosp Disaster Med. 2023 Aug;38(4):546-547. doi: 10.1017/S1049023X2300599X. Epub 2023 Jul 5. PMID 37403461
- [Background] Matthew J, Mike L, Huang HC, Wang CH, Shih CY, Chen YC, Chiu HY. Effects of personalized music intervention on nurse burnout: A feasibility randomized controlled trial. Nurs Health Sci. 2022 Dec;24(4):836-844. doi: 10.1111/nhs.12984. Epub 2022 Oct 9. PMID 36089738
- [Background] Kacem I, Kahloul M, El Arem S, Ayachi S, Hafsia M, Maoua M, Ben Othmane M, El Maalel O, Hmida W, Bouallague O, Ben Abdessalem K, Naija W, Mrizek N. Effects of music therapy on occupational stress and burn-out risk of operating room staff. Libyan J Med. 2020 Dec;15(1):1768024. doi: 10.1080/19932820.2020.1768024. PMID 32449482